CLINICAL TRIAL: NCT04369352
Title: Non-interventional, Multicenter, Prospective Register Study to Describe the Treatment Pattern of Platinum-sensitive Relapsed Epithelial Ovarian Cancer (ROC) Patients in Austria
Brief Title: Register to Describe the Treatment Pattern of Platinum-sensitive Relapsed Epithelial Ovarian Cancer Patients in Austria
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: AGO R03 ROC
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Recurrent Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Various treatment options exist for patients with platinum-sensitive relapsed epithelial ovarian cancer (ROC).

The register will provide an overview of chosen treatments including the reasons, why these options were chosen.

DETAILED DESCRIPTION:
Patients at their first platinum-sensitive ROC will be invited to participate in the register.

These are all patients with recurrent disease 6 or more months after the last cycle of platinum containing chemotherapy.

The Observation Period will begin by signing the Informed Consent Form (ICF) and will continue for up to a total of 24 months (+/- 4 weeks) after the diagnosis of the first relapse or until patient discontinuation for any reason, or patient's death.

Data on First Study Visit, Subsequent Recurrence during Observation Period and Last Observation will be collected in the electronic Case Report Form (eCRF).

The register will identify symptoms and factors that led to the diagnosis, chosen therapy and the reason for choosing the therapy. At inclusion, data on general patient information, primary diagnosis, previous therapy, and tumor characteristics are collected. During the course of observation data on systemic and maintenance treatments, radiotherapies, surgeries, and outcome are documented.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older
* Presence of first platinum-sensitive ROC (ovarian, peritoneal and/or fallopian tube cancer)
* Must have received at least 4 cycles of chemotherapy during primary therapy
* At time of inclusion a treatment for ROC must be planned
* Patients must not have more than 1 prior line of chemotherapy
* Signed informed consent

Exclusion Criteria:

* No knowledge of spoken and written German
* Signed informed consent is not given

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at their first platinum-sensitive ROC treated within gynecological oncology centers in Austria participating in the register.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-08-09 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
To assess treatment patterns and the reasons for selecting these treatments in patients with platinum-sensitive ROC after first relapse in Austria | Two years
  Descriptive Data Analysis

SECONDARY OUTCOMES:
Progression Free Survival | 2 years per patient
  after first relapse and second relapse, evaluated by clinical practice in each center
Overall Survival | 2 years per patient
  at 24 months
Assess Treatments | 2 years per patient
  treatment duration, number of cycle, treatment exposure, time to next treatment
Overall Survival Description | 2 years per patient
  died due to disease, died due to other reasons, alive

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Hefler, Prim. Dr., Principal Investigator — Ordensklinikum Linz
Locations (9):
- Austria (9):
  - Medical University Graz, Graz
  - Medical University Innsbruck, Innsbruck
  - Bezirkskrankenhaus Kufstein, Kufstein
  - LKH Hochsteiermark, Leoben
  - Bezirkskrankenhaus Lienz, Lienz
  - Kepler Universitätsklinikum Linz, Linz
  - Ordensklinikum Linz, Linz
  - Krankenhaus der Barmherzigen Schwestern Ried, Ried im Innkreis
  - Medical University Vienna, Vienna